CLINICAL TRIAL: NCT04399005
Title: The Efficacy Comparing Daily and After-each-case Room Disinfection in the Endoscopy Unit During the COVID-19 Pandemic.
Brief Title: The Efficacy Comparing Daily and After-each-case Room Disinfection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DACD-HuY-2005
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-05

CONDITIONS: Daily Room Disinfection; After-each-case Room Disinfection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- daily room disinfection (Experimental): Room disinfection was defined as the cleansing and disinfection of the surface of the facility, endoscopist's gown, and air in the endoscopy room after the examination. Specifically, sanitizing wipes wiped the surface of the facility one by one, containing quaternary ammonium salt, alcohol, and interfacial activator; the air disinfection machine continued for 30min of air disinfection. Daily room disinfection was defined as disinfection after completing 8 non-general anesthesia gastroscopy or 4 general anesthesia gastroscopy.
  Interventions: Other: daily room disinfection
- after-each-case room disinfection (Experimental): Room disinfection was defined as the cleansing and disinfection of the surface of the facility, endoscopist's gown, and air in the endoscopy room after the examination. Specifically, sanitizing wipes wiped the surface of the facility one by one, containing quaternary ammonium salt, alcohol, and interfacial activator; the air disinfection machine continued for 30min of air disinfection. After-each-case room disinfection was defined as after completing each case.
  Interventions: Other: after-each-case room disinfection

INTERVENTIONS:
Other: after-each-case room disinfection — After-each-case room disinfection was defined as after completing each case.
  Arms: after-each-case room disinfection
Other: daily room disinfection — Daily room disinfection was defined as disinfection after completing 8 non-general anesthesia gastroscopy or 4 general anesthesia gastroscopy.
  Arms: daily room disinfection

SUMMARY:
The aim of our study was to evaluate the difference of effectiveness between daily and after-each-case room disinfection in the endoscopy unit during the COVID-19 pandemic.

DETAILED DESCRIPTION:
This study divided into 2 groups: daily room disinfection and after-each-case room disinfection. Each group was also subdivided into general anesthesia or non-general anesthesia gastroscopy, and with or without ventilation consultation room.

Samples collection include: operation unit air (six-stage sieve percussion air sampler for sampling, airflow rate 28.3L/min, sampling time 4 min); workstation's mouse (wiping sterile cotton for sampling); endoscopist's gown, control panel buttons, and patient's bed headboard (contact plate for sampling).

ELIGIBILITY:
Inclusion Criteria:

* All the cases received gastroscopy.

Exclusion Criteria:

* High-risk personal through contact history, symptoms, body temperature, COVID-19 virus nucleic acid testing and chest computed tomography (CT) scan.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Qualified rate of room disinfection | 48 hours
  The samples of workstation's mouse, control panel buttons and patient's bed headboard greater than 10 CFU/cm2, samples of endoscopist's gown greater than 200 CFU/suit, and samples of operation unit air greater than 500 CFU/m3 are deemed as an unacceptable level of bioburden.
The number of colony-forming units (CFU) | 48 hours
  The number of colony-forming units (CFU) of operation unit air, workstation's mouse, endoscopist's gown, control panel buttons, and patient's bed headboard.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Lu, Principal Investigator — First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data sharing will be consider after study

REFERENCES:
- [Derived] Jin B, Hu Y, Huang L, Cheng X, Zhao J, Yang X, Sun X, Gan T, Lu B. Effectiveness Between Daily and After-Each-Case Room Disinfection of the Endoscopy Unit. Front Public Health. 2021 Oct 5;9:700041. doi: 10.3389/fpubh.2021.700041. eCollection 2021. PMID 34676191

DOCUMENTS (1):
  • Study Protocol (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT04399005/Prot_000.pdf